CLINICAL TRIAL: NCT01480843
Title: Simplification of Diabetes Regimen in Elderly Patients Using Glargine
Brief Title: Simplified Insulin Protocol Using Lantus in Elderly
Acronym: SIMPLE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Joslin Diabetes Center (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011-05
Record Dates: First submitted 2011-11-09; First posted 2011-11-29 (Estimated); Results first posted 2017-11-08 (Actual); Last update posted 2017-11-08 (Actual); Status verified 2017-10

CONDITIONS: Diabetes
Keywords: simplification; glargine; elderly
MeSH Terms: conditions — Diabetes Mellitus | interventions — Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Glargine (Experimental): We plan to add long acting insulin glargine with/without oral medications to the regimen in all patients.
  Interventions: Drug: Glargine

INTERVENTIONS:
Drug: Glargine — Use of glargine with/without other glucose lowering agent to simplify insulin regimen in older adults
  Other Names: Lantus

SUMMARY:
The purpose of this study is to find out if simplifying your diabetes treatment by decreasing number of insulin injections, with the help of a long acting insulin called glargine, can decrease the episodes of low blood glucose.

DETAILED DESCRIPTION:
As patients with diabetes age, adverse social and medical problems may arise. Because of these problems patients, even those managing their diabetes for many years, find it difficult to continue with complicated insulin schedules. This may lead to errors in treatment and poor glucose control. Simplification of treatment has been found to the decrease risk of low blood glucose, a very dangerous condition at this age. In a previous study, the investigators found that simplifying treatment did not cause the blood sugars to rise out of control. In this study, the investigators plan to simplify insulin treatment and monitor for low glucose episodes with help of a continuous glucose monitor and A1C (measure of average glucose control over 3 months). The investigators will simplify the treatment by adding glucose lowering medications that you can take by mouth, in addition to the injection of long acting insulin called glargine.

ELIGIBILITY:
Inclusion Criteria:

* Age 70 years or older
* Diagnosis of diabetes mellitus Type II
* At least 2 (short-acting or mixed) insulin injections per day
* At least 1 episode of hypoglycemia (glucose value <70) on screening CGM

Exclusion Criteria:

* Patients with the following illnesses in the past 12 months Myocardial infarction Angina Coronary artery bypass grafting Percutaneous transluminal coronary angiography Cerebrovascular event (stroke, TIA)
* Active liver disease (history of cirrhosis or LFT > 3 times normal)
* On dialysis or with severe renal dysfunction (creatinine clearance <20 ml/min)
* Malignancy that limits life span to less than 18 months
* Patients seen in the geriatric clinic who already have simplified regimen as proposed in the study

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 65 (Actual)
Dates: Start 2011-06; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medha N Munshi, MD, Principal Investigator — Joslin Diabetes Center
Locations (1):
- Joslin Diabetes Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Narayan KM, Boyle JP, Geiss LS, Saaddine JB, Thompson TJ. Impact of recent increase in incidence on future diabetes burden: U.S., 2005-2050. Diabetes Care. 2006 Sep;29(9):2114-6. doi: 10.2337/dc06-1136. No abstract available. PMID 16936162
- [Background] Economic consequences of diabetes mellitus in the U.S. in 1997. American Diabetes Association. Diabetes Care. 1998 Feb;21(2):296-309. doi: 10.2337/diacare.21.2.296. PMID 9539999
- [Background] Bertoni AG, Kirk JK, Goff DC Jr, Wagenknecht LE. Excess mortality related to diabetes mellitus in elderly Medicare beneficiaries. Ann Epidemiol. 2004 May;14(5):362-7. doi: 10.1016/j.annepidem.2003.09.004. PMID 15177276
- [Background] Blaum CS, Ofstedal MB, Langa KM, Wray LA. Functional status and health outcomes in older americans with diabetes mellitus. J Am Geriatr Soc. 2003 Jun;51(6):745-53. doi: 10.1046/j.1365-2389.2003.51256.x. PMID 12757559
- [Background] Bonsignore P DL, Suhl E, Sternthal A, Giusti J, Munshi MN. Unrecognized Errors in Insulin Injection Techniques Are Frequent in Older Adults Even with Longer Duration of Insulin Use. In: American Diabetes Association annual meeting 2009; 2009; New Orleans LA; 2009. p. 913-P.
- [Background] Medha N. Munshi EB, Ramachandiran Cooppan. Diabetes in the Older Adult. In: Richard S. Beaser MatSoJDC, ed. Joslin's Diabetes Deskbook : A guide for primary care providers. 2nd ed. Boston: Joslin Diabetes Center; 2007:623-38.
- [Background] Shorr RI, Ray WA, Daugherty JR, Griffin MR. Incidence and risk factors for serious hypoglycemia in older persons using insulin or sulfonylureas. Arch Intern Med. 1997 Aug 11-25;157(15):1681-6. PMID 9250229
- [Background] McAulay V FB. Hypoglycemia in diabetes in old age. In: Sinclair A, Finucane P, ed. 2nd ed. Chichester, UK: John wiley and sons; 2001:133-52.
- [Background] Desouza C, Salazar H, Cheong B, Murgo J, Fonseca V. Association of hypoglycemia and cardiac ischemia: a study based on continuous monitoring. Diabetes Care. 2003 May;26(5):1485-9. doi: 10.2337/diacare.26.5.1485. PMID 12716809
- [Background] Frier BM. Hypoglycaemic valleys: an under-recognised problem in type 2 diabetes? Int J Clin Pract Suppl. 2002 Jul;(129):12-9. PMID 12166599
- [Background] Zammitt NN, Frier BM. Hypoglycemia in type 2 diabetes: pathophysiology, frequency, and effects of different treatment modalities. Diabetes Care. 2005 Dec;28(12):2948-61. doi: 10.2337/diacare.28.12.2948. No abstract available. PMID 16306561
- [Background] Ayres D SE, Capelson R, Weinger K, Munshi M. Identifying Barriers to Diabetes Education and Self-Care in Older Adults. In: American diabetes Association 65th scientific sessions 2005; San Diego CA; 2005. p. 941-P
- [Background] Munshi M, Grande L, Hayes M, Ayres D, Suhl E, Capelson R, Lin S, Milberg W, Weinger K. Cognitive dysfunction is associated with poor diabetes control in older adults. Diabetes Care. 2006 Aug;29(8):1794-9. doi: 10.2337/dc06-0506. PMID 16873782
- [Background] Munshi MN DL, Iwata I, Suhl E, Giusti J, Bonsignore P, Sternthal A The Risk of Hypoglycemia Is a Treatment-Limiting Factor in Older Adults Even with Poor Glycemic Control. In: American Diabetes Association annual meeting 2009; 2009; New Orleans LA; 2009. p. 2123-PO.
- [Background] Munshi MN, Hayes M, Sternthal A, Ayres D. Use of serum c-peptide level to simplify diabetes treatment regimens in older adults. Am J Med. 2009 Apr;122(4):395-7. doi: 10.1016/j.amjmed.2008.12.008. PMID 19332236
- [Background] Kovatchev BP, Clarke WL, Breton M, Brayman K, McCall A. Quantifying temporal glucose variability in diabetes via continuous glucose monitoring: mathematical methods and clinical application. Diabetes Technol Ther. 2005 Dec;7(6):849-62. doi: 10.1089/dia.2005.7.849. PMID 16386091
- [Background] Hendriksen C, Faber OK, Drejer J, Binder C. Prevalence of residual B-cell function in insulin-treated diabetics evaluated by the plasma C-etide response to intravenous glucagon. Diabetologia. 1977 Dec;13(6):615-9. doi: 10.1007/BF01236316. PMID 338408
- [Background] Faber OK, Binder C. C-peptide response to glucagon. A test for the residual beta-cell function in diabetes mellitus. Diabetes. 1977 Jul;26(7):605-10. doi: 10.2337/diab.26.7.605. PMID 326604
- [Background] Montorio I, Izal M. The Geriatric Depression Scale: a review of its development and utility. Int Psychogeriatr. 1996 Spring;8(1):103-12. doi: 10.1017/s1041610296002505. PMID 8805091
- [Background] Arbuthnott K, Frank J. Trail making test, part B as a measure of executive control: validation using a set-switching paradigm. J Clin Exp Neuropsychol. 2000 Aug;22(4):518-28. doi: 10.1076/1380-3395(200008)22:4;1-0;FT518. PMID 10923061
- [Background] Welch G, Weinger K, Anderson B, Polonsky WH. Responsiveness of the Problem Areas In Diabetes (PAID) questionnaire. Diabet Med. 2003 Jan;20(1):69-72. doi: 10.1046/j.1464-5491.2003.00832.x. PMID 12519323
- [Background] Polonsky WH, Anderson BJ, Lohrer PA, Welch G, Jacobson AM, Aponte JE, Schwartz CE. Assessment of diabetes-related distress. Diabetes Care. 1995 Jun;18(6):754-60. doi: 10.2337/diacare.18.6.754. PMID 7555499
- [Background] Jacobson AM, de Groot M, Samson JA. The evaluation of two measures of quality of life in patients with type I and type II diabetes. Diabetes Care. 1994 Apr;17(4):267-74. doi: 10.2337/diacare.17.4.267. PMID 8026281
- [Background] Weinger K, Butler HA, Welch GW, La Greca AM. Measuring diabetes self-care: a psychometric analysis of the Self-Care Inventory-Revised with adults. Diabetes Care. 2005 Jun;28(6):1346-52. doi: 10.2337/diacare.28.6.1346. PMID 15920050

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Glargine
Started | 65
Completed | 60
Not Completed | 5

BASELINE CHARACTERISTICS:
Arm/Group | Glargine
Number analyzed (Participants) | 65
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 65
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32
  Male | 33
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 11
  White | 54
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 65

OUTCOME MEASURES:

1. Primary Outcome: Change in Duration of Hypoglycemia Episodes
Description: duration of hypoglycemia measured by continuous glucose monitoring
Time Frame: baseline, 5 months, 8 months
Population: Subject drop outs
Measure: Mean (Standard Deviation); unit: minutes of hypoglycemia
Arm/Group | Glargine
Number analyzed (Participants) | 65
minutes of hypoglycemia
  Baseline | 277 (252)
  5 months: number analyzed (Participants) | 60
  5 months | 111 (184)
  8 months: number analyzed (Participants) | 58
  8 months | 97 (163)

2. Primary Outcome: Change in Frequency of Hypoglycemia Episodes From Baseline, 5 Months, 8 Months
Description: frequency of hypoglycemia episodes measured by continuous glucose monitoring per 5 days of continuous glucose monitoring data
Time Frame: baseline, 5 months, 8 months
Population: Subject drop outs
Measure: Mean (Standard Deviation); unit: episodes of hypoglycemia
Arm/Group | Glargine
Number analyzed (Participants) | 65
episodes of hypoglycemia
  Baseline | 4.3 (3.0)
  5 months | 1.8 (2.0)
  8 months | 1.5 (2.0)

ADVERSE EVENTS:
Time Frame: Adverse Event data was collected during the 8 month time period that the participants were in the trail.
Description: Participants were contacted ona weekly or bi-weekly basis to discuss blood glucose readings and an other issues that they had been having.
Arm/Group | Glargine
All-Cause Mortality (participants affected / at risk) | 3/65
Serious Adverse Events (participants affected / at risk) | 18/65
Other Adverse Events (participants affected / at risk) | 4/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Glargine (N=65)
Death (General disorders) | 3 (3) — Subject passed away from unknown causes
Bowel Obstruction (Gastrointestinal disorders) | 1 (1) — Subject hospitalized for bowel obstruction.
hysterectomy (Reproductive system and breast disorders) | 1 (1) — subject hospitalized for hysterectomy
Stroke (Vascular disorders) | 3 (3) — 2 subjects had strokes and subsequent hospitalization, unrelated to study intervention.
Hospitalization for gout (General disorders) | 1 (2) — subject hospitalized for gout flare up, unrelated to study intervention.
Cardiac stent placed (Cardiac disorders) | 3 (3) — Subject hospitalized for cardiac stent placement. Unrelated to study intervention.
Hospitalization for internal bleeding (General disorders) | 2 (3) — Subject hospitalized due to internal bleeding from mediation unrelated to study intervention.
Hospitalization for Cellulitis (Infections and infestations) | 1 (1) — subject hospitalized for cellulitis unrelated to study intervention.
Hospitalization due to fall (General disorders) | 1 (1) — Subject tripped and fell, resulting in hospitalization. Unrelated to study procedures.
Hospitalization for Acute renal failure (Renal and urinary disorders) | 2 (2) — hospitalization for acute on chronic renal failure, thought to be interstitial nephritis. Unrelated to study intervention
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Glargine (N=65)
Prednisone Taper Needed (General disorders) | 4 (6) — Subjects paused their time in the study due to the use of prednisone, unrelated to study intervention. Prednisone affected blood glucose readings during this time.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No